CLINICAL TRIAL: NCT02691559
Title: The Possible Effect Of Amniotic Fluid pH On Neonatal Morbidities In Maternal Inflammation/Infection Associated Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seda Yilmaz Semerci, Fellowship of Neonatology, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2016-02-01; First posted 2016-02-25 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Distress Syndrome; Transient Tachypnea of Newborn; Intrauterine Growth Retardation
MeSH Terms: conditions — Respiratory Distress Syndrome; Transient Tachypnea of the Newborn; Fetal Growth Retardation

ARMS (2):
- maternal inflammation group (Active Comparator): Amniotic fluid analysis by blood gas device: evaluate the possible association between maternal inflammation and amniotic fluid pH two groups will be designed. One group will consist of infants born to mothers with infection/inflammation whereas the control group will consist of infants born to mothers without infection/inflammation. In all deliveries amniotic fluid will be taken and will be analyzed by blood gas device.
  Interventions: Device: Amniotic fluid analysis by blood gas device
- normal pregnancy group (Active Comparator): Amniotic fluid analysis by blood gas device: The control group will consist of infants born to mothers without infection/inflammation. In all deliveries amniotic fluid will be taken and will be analyzed by blood gas device.
  Interventions: Device: Amniotic fluid analysis by blood gas device

INTERVENTIONS:
Device: Amniotic fluid analysis by blood gas device — Amniotic fluid analysis by blood gas device in maternal inflammation group vs normal pregnancy group

SUMMARY:
Amniotic fluid (AF) pH can be affected by the maternal and/or fetal conditions such as PPROM, prematurity or fetal distress. It is known that fetal urine is the major content of AF since 20th gestational week. Besides fetal alveolar fluid (FAF), gastrointestinal tract, umbilical cord and fetal side of placenta are important sources for AF. Bombesin-like peptides, 8-hydroxydeoxyguanosine in fetal urine and leukotriene E(4), lecithin, sphingomyelin, lamellar body in FAF are molecules acting on fetal lung maturation. Varying levels of these molecules relevant to the stage of lung maturation may constitute an association to AF pHTo detect the possible effect of AF pH on neonatal respiratory morbidities 1 milliliters of AF is aspirated during C-section before incision of membranes. pH value of AFs were analyzed by the blood gas machine (Siemens RAPIDLab®1200 Systems) of NICU. Maternal and neonatal demographic features and clinical outcomes, incidences of morbidities such as respiratory distress syndrome (RDS), transient tachypnea of the newborn (TTN) are all recorded.

ELIGIBILITY:
Inclusion Criteria:

Inflammation/infection associated pregnancies Normal healthy pregnancies

Exclusion Criteria:

Congenital abnormalities Chromosomal abnormalities Blood contaminated amniotic fluid

Max Age: 5 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
A total of 200 amniotic fluid (1ml per one) would be collected and analyzed for the study. | through study completion, an average of 8 months
  Amniotic fluid will be analysed for the value of its pH
A total of 200 amniotic fluid (1ml per one) would be collected and analyzed for the study. | through study completion, an average of 8 months
  Amniotic fluid will be analysed for the value of its contents of electrolytes such as sodium, potassium, chlorid.

SECONDARY OUTCOMES:
A total of 200 amniotic fluid (1ml per one) would be collected and analyzed for the study. | through study completion, an average of 8 months
  Amniotic fluid will be analyzed for primary outcome measures by conventional methods and devices.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yilmaz Semerci, MD, Principal Investigator — Postdoctoral Fellow of Neonatology
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No